CLINICAL TRIAL: NCT05568641
Title: Immunohistochemical Expression of Vitamin-D Receptor in Laryngeal Squamous Cell Carcinoma
Brief Title: Vitamin-D Receptor in Laryngeal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Abdelnaby, Lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-22-09-12
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Laryngeal Carcinoma
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laryngeal squamous cell carcinoma (LSCC) is the second most common primary malignant tumor of the respiratory tract after lung cancer and the second most common primary epithelial malignant tumor of the head and neck. The age of onset of LSCC is mostly between 50 and 70 years, with a male to female ratio of approximately 4:1 .According to estimates by the American Cancer Society, in the United States, approximately 12,470 new cases of laryngeal cancer will be diagnosed and 3,820 people will die from laryngeal cancer in 2022.

The nuclear vitamin D receptor (VDR) is involved in multiple pathways that have many points of convergence. Some of these pathways are implicated in carcinogenesis thus the suggestion that VDR has a role to play in the biology of cancer [3]. Recent evidence indicates that the active form of vitamin D (1alpha, 25-dihydroxycholecalciferol) (VD) exhibits several different effects on normal and cancerous cells, including up-regulation of anti- proliferation and pro-apoptotic factors, as well as inhibition of cell-cycle promoters and growth factor signaling pathways. Thus it is useful as an anti-neoplastic agent in several human malignancies.

Studies in cell and animal model systems, as well as clinical trials have recognized the potential usefulness of VD and VD analogues as agents that enhance the anti-proliferative/cytotoxic effects of chemotherapy and ionizing radiation. Thus, at concentrations that produce limited hypercalcemia, these agents may be used as adjuncts to conventional chemotherapy and radiotherapy. We aim to analyze the expression of VDR in LSCC to determine potential for active VD therapy in such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Both endoscopic and excisional biopsy specimens.
2. All the studied cases include sufficient materials for the immunohistochemical study.
3. Complete clinical data

Exclusion Criteria:

1. Patients with recurrence of the primary tumor.
2. Patients with a history of preoperative chemotherapy and/or radiotherapy.
3. Insufficient or tiny tissue biopsies

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study will be carried out on 50 LSCC specimens that were collected randomly from archives of Pathology Department, Faculty of Medicine, Sohag University
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and prognosis of laryngeal squamous cell carcinoma | Two or three days after staining tissue sections with Vit D receptor antibody
  Immunohistochemical Expression of Vitamin-D Receptor in Laryngeal Squamous Cell Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Abdelnaby, Lecturer, Principal Investigator — Faculty of medicine ,Sohag university

IPD SHARING:
Plan to Share IPD: Undecided